CLINICAL TRIAL: NCT02103049
Title: The Impact of Ezetimibe on Biochemical Markers of Cardiovascular Risk in Kidney Transplant Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Gregor Mlinsek, MD PhD, University Medical Centre Ljubljana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCL-2014-TX
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Dyslipidemia; Transplants
MeSH Terms: conditions — Dyslipidemias | interventions — Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ezetimibe, dyslipidemia, kidney transplant (Other)
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Ezetimibe — Patients on standard immunosuppressive therapy with statin will be added ezetimibe for 6 months. Thereafter ezetimibe will be discontinued for three months. Biochemical parameters will be analysed at the time of enrolment, after 3 months, 6 months and 9 months.

SUMMARY:
In kidney transplant patients atherosclerosis process is accelerated even in asymptomatic patients. This is mainly the consequence of immunosuppressive therapy. Dyslipidemia is treated with statins in low doses only as high doses can lead to rhabdomyolysis and are therefore contraindicated. As second lipid lowering agent most commonly ezetimibe is used. The investigators hypothesise that ezetimibe as a second lipid lowering drug in kidney transplant patients lowers LDL cholesterol for additional 10 per cent.

DETAILED DESCRIPTION:
In addition to observing the lipid profile the investigators intend to look for other pathophysiological effects of ezetimibe, such as its influence on oxidative stress, endothelial function and inflammatory biochemical markers.

ELIGIBILITY:
Inclusion Criteria:

LDL > 2.5 mM, Already treated with statin, Stable renal function of various GFR, Men or women older than 18 years, Signed informed consent.

Exclusion Criteria:

Acute heart disease or any heart disease in the last 3 months, kidney graft failure, active systemic inflammatory disease, active malignant disease, chronic diarrhea and malabsorption, transaminases increased > 3 fold, creatin kinase increased > 5 fold, hypersensitivity reactions, active peptic ulcer disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Decrease of LDL cholesterol concentration. | At enrolment, at three, six and nine months thereafter.
  The investigators expect the LDL cholesterol concentration to lower for at least 10%.

SECONDARY OUTCOMES:
Change in oxidative markers | At enrolment, at three, six and nine months thereafter.
  Change in oxidative markers, inflammation and endothelial function.

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Mlinsek, MD, PhD, Principal Investigator — University Medical Center Ljubljana, Slovenia
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia, Slovenia